CLINICAL TRIAL: NCT00323778
Title: Prospective Assessment of the Efficacy of Intra-Articular Hyaluronate to Affect Extracellular Matrix Changes in Patients With Osteoarthritis
Brief Title: Prospective Assessment of the Efficacy of Hyaluronate Knee Injections in Patients With Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Lisa A. Mandl MD MPH, Hospital for Special Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 25107
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Knee Osteoarthritis
Keywords: hyalgan; knee; osteoarthritis; MRI
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Hyaluronic Acid

INTERVENTIONS:
Drug: Hyalgan

SUMMARY:
This study looks at the effect of an injectable medication called Hyalgan on the cartilage of the knee in people who have osteoarthritis ("wear and tear arthritis") of the knee. Hyalgan is a medication which is injected into the knee, and is FDA approved to treat knee arthritis. We will be using magnetic resonance imaging (MRI) and x-rays to look at knee cartilage to see how it responds over the course of a year to the injections. A comparison to patients taking oral pain medication will be made.

ELIGIBILITY:
Inclusion Criteria:

* age 45-90
* seeking medical care for painful knee osteoarthritis
* alignment based on AP standing radiographs of neutral to 10º of valgus
* no prior surgery on the ipsilateral knee
* no history of major trauma to either knee or either hip
* no history of congenital hip dysplasia
* No history of inflammatory synovitis or crystalline arthropathy
* No history of systemic rheumatic disease
* cruciate and collateral ligament stability, defined by clinical examination
* meniscus intact (MRI grade II degenerative signal acceptable)
* Noyes compartment score: no greater than 50% of cartilage thickness over an area greater than 15mm
* If bilateral OA, the most painful knee, (as documented by VAS scale for pain) which qualifies for the study will be entered.
* If taking glucosamine chondroitin sulfate, discontinue at least one month prior to HA injections

Exclusion Criteria:

* previous IA HA injection in the ipsilateral knee
* IA steroid in the ipsilateral knee in the past 3 months
* MR evidence of inflammatory or hypertrophic synovitis
* Large joint effusion with a ballotable patella on baseline clinical exam
* Inability to safely perform MR imaging
* Active systemic infection
* Active malignancy (except non-melanomatous skin cancer)
* Allergies to HA or chicken products
* Clinical symptoms of an acute meniscal tear (locking, new acute mechanical symptoms etc…)
* A recent injury to the knee
* Radiographic evidence of Grade III or IV Kellgren and Lawrence OA
* Chondrocalcinosis on radiographs
* Unwilling to discontinue or avoid glucosamine chondroitin sulfate for the 12 month study period
* People taking blood thinners or who have bleeding problems
* Anticipated lower extremity surgery during the next 12 months
* BMI >30 kg/m2

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Mandl, MD MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States